CLINICAL TRIAL: NCT05689866
Title: Study of Bladder-sphincter Symptoms in Functional Neurological Disorders
Acronym: URO-TNF
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221001
Record Dates: First submitted 2022-11-14; First posted 2023-01-19 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-06

CONDITIONS: Urinary Bladder Sphincter Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A significant proportion of patients with functional neurological disorders (FND) report urinary, anorectal or genitosexual disorders. However, until now, no study has focused on bladder-sphincter disorders in patients with FND. The symptoms of this pathology are, therefore, not precisely characterized.

Thus, the objective of this research is to specify if urinary, anorectal or sexual disorders can be observed in patients suffering from functional neurological disorders and to better describe them in order to propose better therapeutic options.

DETAILED DESCRIPTION:
In this clinical study the investigators want to prospectively include all patients presenting to a neurology consultation or day hospital for management of a motor or sensory FND.The patients will first be evaluated for their sphincter functions by self questionnaires. For those where a vesico-sphincter complaint is demonstrated, a neuro-urological consultation will be proposed. A follow-up will then be done, if necessary, in neurology and neuro-urology.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Diagnosis of Functional Neurological Disorders according to DSM 5 criteria
* No neurological comorbidity that could account for the sphincter disorders
* Normal cerebral and spinal cord magnetic resonance imaging.
* Patient affiliated to a French social security system
* Patient informed and not objecting to participate in the study

Non inclusion Criteria :

* Presence of neurological comorbidity that can account for sphincter disorders (e.g. multiple sclerosis, chronic neuropathy, etc.)
* Pregnancy in progress
* Candidate for surgery or locoregional treatment
* Patient subject to legal protection measures.
* Patient under state medical assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to a neurology consultation or day hospital for management of a functional motor or sensory disorder.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
presence of at least one bladder-sphincter disorder | inclusion
  This primary endpoint will be measured by the score of the questionnairies which will define the presence of a vesicosphincter disorder (USP), anorectal disorder (Kess and Wexner) or sexual genital disorder (FSFI/IIEF5)

SECONDARY OUTCOMES:
evaluate the nature of bladder and bowel disorders in patients with NFT | inclusion
  the score of the different questionnairies vesicosphincter disorder (USP), anorectal disorder (Kess and Wexner) or sexual genital disorder (FSFI/IIEF5) that will define the presence of a bladder symptoms
Assess the persistence of bladder and sphincter complaints in patients with NFTs | 24months
  the score of the questionnairies vesicosphincter disorder (USP), anorectal disorder (Kess and Wexner) or sexual genital disorder (FSFI/IIEF5) that will define the presence of a bladder symptoms
Evaluate whether patients with significant vesico-sphincter complaints differ from patients without complaints, including demographic, traumatic, and NFT semiology. | 24months
  comparison of the characteristics of patients on the vesico-sphincter level
To assess whether the clinical and paraclinical patterns of bladder and sphincter disorders differ according to the type of NFT. | 24months
  Analysis of urodynamic assessment data

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Avicenne-Neurology, Bobigny, France